CLINICAL TRIAL: NCT03151278
Title: Multi-center, Randomized, Controlled Trial to Compare Feasibility, Safety and Efficacy of Zero-Fluoroscopic Navigation With Conventional Fluoroscopic Navigation for the Ablation of Right Atrial Arrhythmias
Brief Title: Zero Fluoroscopic Ablation Versus Conventional Fluoroscopic Ablation for Right Atrial Arrhythmias
Acronym: ZFA-RAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Xinyang Central Hospital (Other); Ningbo No. 1 Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); First Affiliated Hospital of Guangxi Medical University (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Guangdong Provincial People's Hospital (Other); Zhongshan Hospital Xiamen University (Other)
Responsible Party: Principal Investigator, Yan Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHCDD-ZF-RAA-20110131
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Atrial Arrhythmia; Atrial Premature Complexes; Atrial Tachycardia
Keywords: Fluoroscopy; Ablation; Three dimensional; Atrial arrhythmia; Radiation
MeSH Terms: conditions — Atrial Premature Complexes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero-fluoroscopy ablation (Experimental): Atrial arrhythmias will be mapped and ablated under the guidance of three-dimensional mapping system without fluoroscopy.
  Interventions: Procedure: Zero-fluoroscopy ablation
- Conventional fluoroscopy ablation (Active Comparator): Atrial arrhythmias will be mapped and ablated under fluoroscopic guidance plus three-dimensional mapping system.
  Interventions: Procedure: Conventional fluoroscopy ablation

INTERVENTIONS:
Procedure: Zero-fluoroscopy ablation — Catheter ablation will be performed under the guidance of one kind of three-dimensional navigation system and without fluoroscopic guidance.
  Arms: Zero-fluoroscopy ablation
Procedure: Conventional fluoroscopy ablation — Catheter ablation will be performed using fluoroscopy plus one kind of three-dimensional navigation system.
  Arms: Conventional fluoroscopy ablation

SUMMARY:
This study is intended to compare the feasibility, safety and efficacy of a zero-fluoroscopic approach with conventional fluoroscopic approach as performing catheter ablation of right atrial arrhythmias.

DETAILED DESCRIPTION:
Catheter ablation is a well-established treatment to treat patients with a wide range of heart rhythm disturbances.

Fluoroscopy is the imaging modality routinely used for cardiac device implantation and electrophysiological procedures. Due to the rising concern regarding the harmful effects of radiation exposure to both the patients and operation staffs, novel three-dimensional mapping systems such as Ensite NavX have been developed and implemented in electrophysiological procedure for the navigation of catheters inside the heart chambers.

Ensite NavX is a promising system to guide catheters inside the cardiac chambers and vessels without the use of fluoroscopy.

This study is intended to compare the feasibility, safety and efficacy of a zero-fluoroscopic approach with conventional fluoroscopic approach as performing catheter ablation of right atrial arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Atrial Tachycardia
* Atrial Premature Complexes

Exclusion Criteria:

* Left Atrial Premature Complexes
* Left Atrial Tachycardia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Total success rates | 3 months
  The patients have no related arrhythias or recurrence during follow up.

SECONDARY OUTCOMES:
Total procedure time | during procedure
  The patients have no related arrhythias or recurrence during follow up.
Fluoroscopy time | during procedure
  From skin puncture to withdrawal of all the catheters.
Complications | 6 months
  The patients have no related complications during follow up.
Immediate success rate | 24 hours
  Electrophysiologic study shows success of ablation
Recurrence rate | 6 months
  The patients have no related arrhythias or recurrence during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelsomino S, La Meir M, Luca F, Lorusso R, Crudeli E, Vasquez L, Gensini GF, Maessen J. Treatment of lone atrial fibrillation: a look at the past, a view of the present and a glance at the future. Eur J Cardiothorac Surg. 2012 Jun;41(6):1284-94. doi: 10.1093/ejcts/ezr222. Epub 2012 Jan 10. PMID 22233800
- [Background] Birnie D, Healey JS, Krahn AD, Ahmad K, Crystal E, Khaykin Y, Chauhan V, Philippon F, Exner D, Thibault B, Hruczkowski T, Nery P, Keren A, Redfearn D. Prevalence and risk factors for cervical and lumbar spondylosis in interventional electrophysiologists. J Cardiovasc Electrophysiol. 2011 Sep;22(9):957-60. doi: 10.1111/j.1540-8167.2011.02041.x. Epub 2011 Mar 8. PMID 21385267
- [Background] Sra J, Krum D, Hare J, Okerlund D, Thompson H, Vass M, Schweitzer J, Olson E, Foley WD, Akhtar M. Feasibility and validation of registration of three-dimensional left atrial models derived from computed tomography with a noncontact cardiac mapping system. Heart Rhythm. 2005 Jan;2(1):55-63. doi: 10.1016/j.hrthm.2004.10.035. PMID 15851266
- [Background] Oral H, Crawford T, Frederick M, Gadeela N, Wimmer A, Dey S, Sarrazin JF, Kuhne M, Chalfoun N, Wells D, Good E, Jongnarangsin K, Chugh A, Bogun F, Pelosi F Jr, Morady F. Inducibility of paroxysmal atrial fibrillation by isoproterenol and its relation to the mode of onset of atrial fibrillation. J Cardiovasc Electrophysiol. 2008 May;19(5):466-70. doi: 10.1111/j.1540-8167.2007.01089.x. Epub 2008 Feb 4. PMID 18266669
- [Background] Razminia M, Manankil MF, Eryazici PL, Arrieta-Garcia C, Wang T, D'Silva OJ, Lopez CS, Crystal GJ, Khan S, Stancu MM, Turner M, Anthony J, Zheutlin TA, Kehoe RF. Nonfluoroscopic catheter ablation of cardiac arrhythmias in adults: feasibility, safety, and efficacy. J Cardiovasc Electrophysiol. 2012 Oct;23(10):1078-86. doi: 10.1111/j.1540-8167.2012.02344.x. Epub 2012 May 9. PMID 22571735